CLINICAL TRIAL: NCT02285400
Title: Effects of Continuous Positive Airway Pressure (CPAP) Level on Respiratory Mechanics and Central Drive in Patients With Chronic Obstructive Pulmonary Disease
Brief Title: Effects of CPAP Level on Respiratory Mechanics and Central Drive in Patients With COPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zhujiang Hospital (Other)
Collaborators: Guangzhou Institute of Respiratory Disease (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LY20140927
Record Dates: First submitted 2014-10-11; First posted 2014-11-07 (Estimated); Last update posted 2015-12-31 (Estimated); Status verified 2015-07

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: COPD; CPAP; Central Drive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Moderate COPD patients (Experimental): Patients are connected to the noninvasive ventilator and incremental CPAP level is performed.
  Interventions: Procedure: CPAP level
- Severe COPD patients (Experimental): Patients are connected to the noninvasive ventilator and incremental CPAP level is performed.
  Interventions: Procedure: CPAP level

INTERVENTIONS:
Procedure: CPAP level — CPAP level ranges between 4 and 12 cm water column (cmH2O), each pressure increment for 1 cmH2O.

SUMMARY:
Chronic Obstructive Pulmonary Disease (COPD) is a common respiratory disease characterized by airflow limitation that is progressive and not fully reversible. Expiratory flow limitation (EFL) is the main mechanism leading to dynamic pulmonary hyperinflation (DPH) and intrinsic positive end-expiratory pressure (PEEPi). DPH and PEEPi lead to increased inspiratory muscle efforts and impaired central drive mechanical and ventilation coupling, which is an important mechanism of dyspnea. Appropriate setting of extrinsic PEEP (PEEPe) can decrease inspiratory efforts and work of breathing, improve patient-ventilator synchrony in severe COPD patients with PEEPi and treated with mechanical ventilation. Nevertheless, the effects of CPAP/PEEPe level on respiratory mechanics, especially on central drive mechanical and ventilation coupling, still need further investigations.

In the present study, about 40 patients with COPD will be recruited as research subjects. And the investigators aim to observe the changes in respiratory mechanics, central drive mechanics, central drive mechanical and ventilation coupling at different levels of CPAP. Contrast analysis will be conducted to evaluate the effects of CPAP level on respiratory mechanics and central drive during DPH, which may provide a reasonable basis for the clinical application of CPAP to COPD patients and the exploration of a new reasonable CPAP setting method.

DETAILED DESCRIPTION:
Patients with COPD are divided into two groups: moderate group and severe group, both of which are intervented by CPAP level. The static pressure volume curves of the lung and chest wall (Campbell diagram) were established with slow deep respiratory manoeuvre. Before using CPAP level, we will measure the relevant parameters of lung volume, respiratory flow, diaphragm electromyogram, central drive mechanical and ventilation coupling. Then incremental CPAP level will be applied to investigate the effects of CPAP level on the above mentioned respiratory mechanics parameters.

ELIGIBILITY:
Inclusion Criteria:

* Patients from Zhu jiang Hospital,Southern Medical University
* Patients aged 40-70 years old
* Patients with pulmonary function test of forced expiratory volume at one second (FEV1)/forced vital capacity(FVC) < 70% and 30% ≤ FEV1%pred < 80%
* Patients in a clinically stable state
* Patients who signed informed consent.

Exclusion Criteria:

* Patients with signs of an airway infection
* Patients with an acute exacerbation during the previous 4 weeks
* Patients with giant bulla(≥3cm in diameter)
* Patients with recent upper abdominal surgery
* Patients with one or more of the following diseases: esophageal cancer, reflux esophagitis, severe obstructive sleep apnea (apnea hypopnea index>15/hr), neuromuscular disease, or significant heart failure
* Patients with poor compliance.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-11; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Diaphragmatic function | Change from baseline in diaphragm electromyogram at 12 cmH2O CPAP level. (10 minutes later,20minutes later,30 minutes later, 40 minutes later)
  Diaphragmatic function can be assessed by diaphragm electromyogram (EMGdi), which reflect the physiological activity of the diaphragm and indicate functional status of the central drive.

SECONDARY OUTCOMES:
Respiratory pressure | Chang from baseline in respiratory pressure at 12 cmH2O CPAP level.(10 minutes later,20minutes later,30 minutes later, 40 minutes later)
  Respiratory pressure parameters include gastric pressure (Pga), esophageal pressure (Pes), transdiaphragmatic pressure ( Pdi), mouth pressure (Pmo).
Respiratory volume | Chang from baseline in respiratory volume at 12 cmH2O CPAP level. (10 minutes later,20minutes later,30 minutes later, 40 minutes later)
  Respiratory volume is associated with Flow, Inspiratory capacity (IC), tidal volume (VT), respiratory rate (RR), inspiratory time (Ti),expiratory time (Te), minute ventilation (VE).
Degree of dyspnea | Chang from baseline in dyspnea at 12 cmH2O CPAP level. (10 minutes later,20minutes later,30 minutes later, 40 minutes later)
  Difference in the degree of dyspnea can be measured by Borg index.

OTHER OUTCOMES:
Pulse oxygen saturation (SpO2) | Chang from baseline in SpO2 at 12 cmH2O CPAP level. (10 minutes later,20minutes later,30 minutes later, 40 minutes later)
  Change in SpO2 can be recorded by noninvasive monitoring instruments.
End tidal carbon dioxide pressure (PETCO2) | Chang from baseline in PETCO2 at 12 cmH2O CPAP level. (10 minutes later,20minutes later,30 minutes later, 40 minutes later)
  Change in PETCO2 can be recorded by noninvasive monitoring instruments.

CONTACTS AND LOCATIONS:
Overall Officials: Xin Chen, Doctor, Principal Investigator — Zhujiang Hospital,Southern Medical Unversity
Locations (1):
- Zhujiang Hospital,Southern Medical Universtiy, Guangzhou, Guangdong, China